CLINICAL TRIAL: NCT01536860
Title: Glycaemic Response Testing
Brief Title: Glycemic Response Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Reading Scientific Services Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P12-00794
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Glycemic Index; Glycemic Response
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Test Drink (Placebo Comparator): control drink
  Interventions: Other: Dietary Intervention
- Experimental Test Drink 1 (Experimental): control drink containing ingredient 1
  Interventions: Other: Dietary Intervention
- Experimental Test Drink 2 (Experimental): Control drink containing ingredient 2
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — 300 ml of liquid food product
  Arms: Control Test Drink
Other: Dietary Intervention — 300 ml of liquid food product
  Arms: Experimental Test Drink 1
Other: Dietary Intervention — 300 ml of liquid food product
  Arms: Experimental Test Drink 2

SUMMARY:
The purpose of this study is to assess whether added food ingredient(s) affect glycemic responses to a liquid meal tolerance test (LMTT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (not less than 40% males or females
* Non-smoker
* Aged 18 to 55 years
* Have a body mass index between 18.5 to 29.99 kg/m2
* Healthy, non-diabetic, no gastric bypass surgery
* Not allergic to mustard, dairy or soy
* Having a fasting plasma glucose (finger stick) <100 mg/dl (<5.5 mmol/L)
* Willing and able to provide written informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Hart, SCS, Dip, MICR, Principal Investigator — RSSL
Locations (1):
- Reading Scientific Services Limited (RSSL), Reading, Berkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 subjects completed the study. The study was conducted at one clinical research site and study started February, 2012 and was completed in March 2012.
Pre-assignment Details: This was a randomized double blind cross-over study. There was a wash out period of 3 or more days between interventions.
Groups:
- Control Test Drink/Exp Test Drink 1/Exp Test Drink 2: Consume Control Test Drink once over a 15 minute period followed by a 3 day wash out period.
  Consume Exp Test Drink 1 followed by a 3 day wash out period. Consume Exp Test Drink 2 over a 15 minute period
- Exp Test Drink 1/Control Test Drink/Exp Test Drink 2: Consume Exp Test Drink 1 once over a 15 minute period followed by a 3 day wash out period.
  Consume Control Test Drink once over a 15 minute period followed by a 3 day wash out period.
  Consume Exp Test Drink 2 once over a 15 minute period.
- Exp Test Drink 2/Control Test Drink/ Exp Test Drink 1: Consume Exp Test Drink 2 once over a 15 minute period followed by a 3 day wash out period.
  Consume Control Test Drink once over a 15 minute period followed by a 3 day wash out period.
  Consume Exp Test Drink 1 once over a 15 minute period.
Period: First Intervention (1 Day)
Arm/Group | Control Test Drink/Exp Test Drink 1/Exp Test Drink 2 | Exp Test Drink 1/Control Test Drink/Exp Test Drink 2 | Exp Test Drink 2/Control Test Drink/ Exp Test Drink 1
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Washout Period (3 Days)
Arm/Group | Control Test Drink/Exp Test Drink 1/Exp Test Drink 2 | Exp Test Drink 1/Control Test Drink/Exp Test Drink 2 | Exp Test Drink 2/Control Test Drink/ Exp Test Drink 1
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Control Test Drink/Exp Test Drink 1/Exp Test Drink 2 | Exp Test Drink 1/Control Test Drink/Exp Test Drink 2 | Exp Test Drink 2/Control Test Drink/ Exp Test Drink 1
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Washout Period (3 Days)
Arm/Group | Control Test Drink/Exp Test Drink 1/Exp Test Drink 2 | Exp Test Drink 1/Control Test Drink/Exp Test Drink 2 | Exp Test Drink 2/Control Test Drink/ Exp Test Drink 1
Started | 4 | 4 | 4
Completed | 3 | 4 | 4
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Control Test Drink/Exp Test Drink 1/Exp Test Drink 2 | Exp Test Drink 1/Control Test Drink/Exp Test Drink 2 | Exp Test Drink 2/Control Test Drink/ Exp Test Drink 1
Started | 3 | 4 | 4
Completed | 3 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Control Test Drink first, Exp Test Drink 1 first and Exp Test Drink 2 first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Response Measured as the Positive Incremental Area Under the Time-concentration Curve(iAUC) Calculated From Individual Glucose Measurements Upon Consumption of Control and Experimental Test Food Products
Description: The individual glucose measurements were collected at baseline (prior to consumption of each test food product and 15, 30, 45, 60, 90 and 120 minutes following the initiation of consumption of each test food product. The positive incremental area under the time-concentration curve (iAUC) was then calculated for the entire 120 minutes after consumption of each test food product. The results show the differential treatment-related effect on the time-concentration curve (iAUC) for the entire 120 minutes post consumption of each test food product.
Time Frame: 0-120 minutes
Measure: Mean (Standard Error); unit: mmol*min/L
Groups:
- Control Test Drink: Control Drink
  Dietary Intervention : 300 ml of liquid food product
- Experimental Test Drink 1: Control Drink containing ingredient 1
  Dietary Intervention : 300 ml of liquid food product
- Experimental Test Drink 2: Control Drink containing ingredient 2
  Dietary Intervention : 300 ml of liquid food product
Arm/Group | Control Test Drink | Experimental Test Drink 1 | Experimental Test Drink 2
Number analyzed (Participants) | 12 | 12 | 11
mmol*min/L | 100 (17) | 68 (10) | 73 (13)

ADVERSE EVENTS:
Arm/Group | Control Test Drink | Experimental Test Drink 1 | Experimental Test Drink 2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes